CLINICAL TRIAL: NCT01477008
Title: A Prospective, Multi-Center, Randomized Clinical Trial Comparing the Biphasic Cartilage Repair Implant to Marrow Stimulation in the Treatment of Focal Chondral and Osteochondral Lesions of the Knee
Brief Title: BiPhasic Cartilage Repair Implant (BiCRI) IDE Clinical Trial - Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGend Therapeutics Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR09-006; 9907776 (Other: Taiwan FDA - IDE #)
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Chondral or Osteochondral Lesion of Medial Femoral Condyle; Chondral or Osteochondral Lesion of Lateral Femoral Condyle; Chondral or Osteochondral Lesion of Trochlea
Keywords: Knee; Cartilage repair; Cartilage regeneration; Chondral; Osteochondral; Biphasic scaffold; Medical device; Autologous; Synthetic; Medial condyle; Lateral condyle; Trochlea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BiCRI (Experimental): BiPhasic Cartilage Repair Implant
  Interventions: Device: BiPhasic Cartilage Repair Implant
- Marrow Stimulation (Active Comparator): Microfracture or Subchondral Drilling
  Interventions: Procedure: Marrow Stimulation

INTERVENTIONS:
Device: BiPhasic Cartilage Repair Implant — 1 or 2 BiCRI devices, depending on lesion size
  Arms: BiCRI
Procedure: Marrow Stimulation — Microfracture or Subchondral Drilling
  Arms: Marrow Stimulation

SUMMARY:
The purpose of this trial is to evaluate the safety and effectiveness of the Biphasic Cartilage Repair Implant (BiCRI) compared to marrow stimulation in the treatment of chondral and osteochondral lesions located on the medial femoral condyle, lateral femoral condyle, or trochlea of the knee. The hypothesis is that the BiCRI provides an improvement in pain and function as compared to baseline, that is no worse than marrow stimulation at 1 year.

ELIGIBILITY:
Inclusion Criteria

1. Male or female presenting with a single, symptomatic chondral or osteochondral lesion of the medial or lateral femoral condyles or the trochlea requiring primary surgical intervention
2. Skeletally mature (epiphyses are confirmed to be closed on x-ray)
3. ICRS grade 3-4 lesion, Outerbridge grade 4, or OCD grades 3-4
4. Lesion size requires no more than 2 implants (assuming patient were to be randomized to the treatment group). Lesion size will be assessed at the time of the study procedure for all subjects. If the size of the lesion is appropriate for 1 or 2 implants the patient will be randomized. If the lesion is found to be too large the patient will not be included in the trial, but will be treated according to standard of care. Lesion sizes that are considered appropriate include the following:

   * Lesion is 3mm x 3mm or larger and can be completely covered by the small (12.5mm diameter) sizer (excluding small fissures). This lesion should be treated with 1 implant. or
   * Lesion is 3mm x 3mm or larger and cannot be covered by the small sizer, but can be completely covered by the large (oval shaped) sizer (excluding small fissures). This lesion should be treated with 2 implants.
5. Willing and able to refrain from taking pain medications (including: narcotic and non-steroidal anti-inflammatory drugs) for 7 days prior to the baseline preoperative visit and for 7 days prior to the 12-month postoperative visit (i.e., a "wash out" period)
6. Willing and able to return for follow-up over a one year post-operative period
7. Willing and able to comply with all postoperative guidelines

Exclusion Criteria

1. ≥ 55 years old
2. Lesions > grade II on the articular surface of the tibia or patella
3. Kissing lesions (defined as an opposing lesion > grade II on the surface of the tibia or patella). Lesion ≤ grade II on opposing surface would be acceptable.
4. Prior surgical treatment of the lesion
5. Lesion would require more than 2 implants (assuming patient were to be randomized to the treatment group). Lesion sizes that are not considered appropriate include the following:

   * Lesion is smaller than 3mm x 3mm
   * Lesion cannot be completely covered by the large sizer
6. Lesion will require bone grafting
7. Rheumatoid arthritis and other inflammatory arthritis
8. Concomitant comorbidities, such as:

   * ACL instability that will not be corrected before or during the study procedure ("ACL instability" defined as the presence of a positive "pivot shift" test)
   * Significant knee instability that will not be corrected before or during the study procedure
   * Significant malalignment (varus or valgus deformity, patellar malalignment) that will not be corrected before or during the study procedure. Significant malalignment defined as:

     * Any joint space narrowing as compared to the same compartment in the contralateral knee.
     * Mechanical axis alignment outside the tibial spines.
     * Patellofemoral subluxation on sunrise view.
     * History of patellar dislocation or subluxation.
   * Severe meniscal damage ("Severe meniscal damage" defined as > 50% of the meniscus missing or a radial tear extending to the meniscal-synovial junction)
   * Knee stiffness, defined as:

     * Flexion contracture >10°
     * Flexion degree < 115°
9. Body Mass Index (BMI) > 35.0
10. Local or systemic infection, not including asymptomatic urinary tract infection if treated with antibiotics preoperatively
11. Pregnancy or breast feeding
12. Prisoner
13. Patient is involved in a personal litigation (e.g. Worker's Compensation lawsuit) that relates to their knee surgery
14. Patient is actively participating in another medical device, drug, or biologic investigation (active defined as within the last 30 days)
15. Patient otherwise meets the study criteria but refuses to consent in writing to participate in the study

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2011-10; Primary Completion 2019-04 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
IKDC-2000 Subjective Knee Evaluation | 12 months
  Subjective evaluation of knee pain and function (will be captured at preop and each postop visit through 12 months)

SECONDARY OUTCOMES:
IKDC-2000 Knee Examination Form | Preop, 6 weeks, 3 months, 6 months, and 12 months
  Objective evaluation of knee pain and function
IKDC-2000 Current Health Assessment Form | Preop, 6 weeks, 3 months, 6 months, and 12 months
  Subjective evaluation of quality of life (QOL) and activities of daily living (ADL)
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Preop, 6 weeks, 3 months, 6 months, and 12 months
  A subjective instrument to assess the subject's opinion about their knee and associated problems
Pain (VAS): sitting, standing, and squatting | Preop, 6 weeks, 3 months, 6 months, and 12 months
  Subjective evaluation of pain during routine activities
Magnetic Resonance Imagining (MRI) | Preop and 12 months
  MRI to evaluate cartilage and bone condition
Radiographs | Preop, immediate postop, 6 weeks, 3 months, 6 months, 12 months
  Not all views taken at each time frame.
  * Weight bearing full extension AP view (both knees)
  * Rosenberg view (45 degree PA flexion weight bearing, both knees)
  * Lateral view of involved knee
  * Sunrise (skyline) view of involved knee
Adverse Events | Treatment through 12 months
  Documentation of all adverse events from treatment through the end of the study.
Arthroscopy with biopsy | 12 months
  Arthroscopic second look to visualize the repair site. Biopsy of the cartilage and bone region of the treated site. Only performed on patients who agree to second procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Chang, MS, Study Director — BioGend Therapeutics Co.Ltd
Locations (11):
- Taiwan (11):
  - Taipei Medical University-Shuang Ho Hospital, Taipei County, Taipei
  - Show Chwan Memorial Hospital (SCMH), Changhua
  - Chang Gung Memorial Hospital Kaohsiung (CGMH-KS), Kaohsiung City
  - Chang Gung Memorial Hospital Linkou (CGMH-LK), Linkou District
  - China Medical University Hospital (CMUH), Taichung
  - Veterans General Hospital Taichung (VGHTC), Taichung
  - National Cheng Kung University Medical Center (NCKUMC), Tainan
  - National Taiwan University Hospital (NTUH), Taipei
  - Shuang Ho Hospital (SHH), Taipei
  - Taipei Tzu Chi Hospital (TTCH), Taipei
  - Tri-Service General Hospital (TSGH), Taipei

REFERENCES:
- [Derived] Kuo YY, Chiu SQ, Chang WP, Chen CY, Chen CH, Liaw CK, Tan CA, Weng PW. A prospective randomized controlled trial comparing biphasic cartilage repair implant with microfracture in small chondral lesions of knee: findings at five-year-follow-up. J Orthop Surg Res. 2025 Jan 20;20(1):73. doi: 10.1186/s13018-024-05392-6. PMID 39833829
- [Derived] Tseng TH, Chen CP, Jiang CC, Weng PW, Chan YS, Hsu HC, Chiang H. Biphasic cartilage repair implant versus microfracture in the treatment of focal chondral and osteochondral lesions of the knee: a prospective, multi-center, randomized clinical trial. J Orthop Traumatol. 2024 Nov 30;25(1):62. doi: 10.1186/s10195-024-00802-1. PMID 39614986